CLINICAL TRIAL: NCT00274118
Title: DETAIL = Diabetics Exposed to Telmisartan And enalapIL: A Randomised, Double-blind, Parallel-group Comparison of the Renal and Antihypertensive Effects of Telmisartan and Enalapril in Subjects With Mild to Moderate Hypertension and Concurrent Type II Diabetes Mellitus and Diabetic Nephropathy
Brief Title: DETAIL Study: Diabetes Exposed to Telmisartan and Enalapril
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 502.236
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — Telmisartan; Enalapril

INTERVENTIONS:
Drug: telmisartan
Drug: enalapril

SUMMARY:
To compare the renal consequences of two different approaches to blocking the renin angiotensin system in subjects with hypertension and concurrent Type II diabetes mellitus and diabetic nephropathy.

DETAILED DESCRIPTION:
The aims of this study were to compare the renal consequences of two different approaches to blocking the activity of the renin angiotensin system - Angiotensin II antagonism with telmisartan and ACE inhibition with enalapril - in patients with hypertension and concurrent type II diabetes mellitus and diabetic nephropathy.

The study was designed to investigate albumin excretion rates in the short term, and in the longer term, to assess the outcome with respect to maintenance of renal function (GFR) and incidence of clinical endpoints.

Study Hypothesis:

Association of Hypertension and Diabetes Essential hypertension accounts for the majority of hypertension in people with diabetes, particularly in those with type II diabetes, who constitute more than 90% of those with a dual diagnosis of diabetes and hypertension.

Both diabetes and hypertension each confer increased cardiovascular risk, and patients with both conditions have more atherogenic risk factors.

Albumin Excretion as a Therapeutic Marker Microalbuminuria is an early and reliable predictor of diabetic nephropathy in both type I - insulin dependent diabetes mellitus (IDDM) and type II - non insulin dependent diabetes mellitus (NIDDM) patients, nephropathy being characterised by hypertension and an inevitable decline in renal function.

Furthermore, diabetic nephropathy is the single most important cause of end stage renal failure (ESRF) in the western world and over recent years the incidence of ESRF in patients with type II diabetes has dramatically increased.

In addition to predicting nephropathy, in type II diabetes, microalbuminuria also predicts mortality, the major causes of death being related to cardiovascular disease.

Comparison(s):

Selection of an ACE Inhibitor as the Comparative Agent Findings in preclinical studies of animals with diabetes mellitus suggest that ACE inhibitors reduce glomerular damage by one or more mechanisms independent of their antihypertensive effects. Glomerular efferent arteriolar tone is increased in diabetic animals and as a result there is an increase in transcapillary hydraulic pressure. These alterations may decrease the functional integrity of the glomerular capillary wall. In rats with diabetes, the long term administration of an ACE inhibitor diminishes the functional and morphologic evidence of glomerular injury and decreases glomerular transcapillary pressure. Removal of the tonic constrictor effect of angiotensin II on efferent arterioles would be expected to lower glomerular intracapillary pressure while preserving renal plasma flow.

Angiotensin II antagonists appear to be as effective as ACE inhibitors in delaying the progression of renal injury in animal models of diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the ages 35 and 80 years.
2. Current ACE inhibitor therapy for a minimum period of 3 months prior to study entry.
3. Confirmed diagnosis of type II diabetes:

   * Subjects currently treated by diet or diet and oral hypoglycaemic drugs, OR
   * Subjects currently treated with insulin, with a history of onset of diabetes after the age of 40 and a body weight in excess of ideal body weight at the time of diagnosis, and treated with oral agents for a minimum period of two years
4. On treatment diastolic blood pressure of < 95 mmHg.
5. Documentation of a normal renal ultrasound within previous 6 months prior to inclusion (alternate methods eg pyelography, renal isotope method was also acceptable).
6. Mean of three consecutive overnight urinary albumin excretion rates > 20 and < 1000 g/min at the end of the pre-treatment observation period. (A minimum of two of the three samples must be > 20 g/min.)
7. Glycosylated haemoglobin (HbA 1c) < 10%.
8. Serum creatinine < 140 mol/L.
9. Glomerular filtration rate (GFR) > 70 ml/min/1.73 m2.
10. Ability to provide written informed consent.

Exclusion Criteria:

1. Type I diabetes mellitus.
2. Pre-menopausal women (last menstruation < 1 year prior to start of screening period):

   * Who were not surgically sterile (tubal ligation, hysterectomy) or
   * Who were not practising acceptable means of birth control (and do not plan to continue using this method throughout the study). Acceptable methods of birth control include oral, implantable or injectable contraceptives.
   * Who had a positive serum pregnancy test at baseline.
3. Afro-Caribbean subjects.
4. Mean seated SBP > 180 mmHg.
5. Hepatic dysfunction as defined by the following laboratory parameters: SGPT(ALT) or SGOT(AST) > 1.5 times the upper limit of normal.
6. Known causes of renal dysfunction other than diabetic nephropathy.
7. Subjects who had a solitary kidney or known renal artery stenosis.
8. NYHA functional class CHF II - IV.
9. Known drug or alcohol dependency.
10. Subjects receiving any investigational therapy within one month of providing written informed consent.
11. Known hypersensitivity to telmisartan or ACE inhibitors or to any component of the formulation.
12. Subjects with a history of suspected angioedema related to ACE inhibitor therapy.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 1997-07; Primary Completion 2004-01 (Actual); Study Completion 2004-01

PRIMARY OUTCOMES:
Change from baseline in glomerular filtration rate GFR after five years of treatment. | 5 years

SECONDARY OUTCOMES:
Change from baseline in GFR after one, two, three and four years of treatment | Baseline, 1,2,3 and 4 years
Percentage change from baseline in urinary albumin excretion rate | up to 5 years
Change from baseline in creatinine | up to 5 years
Incidence of clinical endpoints (including- end-stage renal disease, myocardial infarction, cerebrovascular accident, congestive heart failure) | up to 5 years
Incidence of all cause mortality | up to 5 years
Changes in vital signs (DBP, SBP, pulse rate) | up to 5 years
Number of patients with Adverse Events | up to 5 years
Physical examination | up to 5 years
Clinical laboratory parameters | up to 5 years
Resting 12-lead ECG | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Ltd./Bracknell
Locations (37):
- Denmark (6):
  - Apopleksiafsnittet, Frederiksberg
  - Boehringer Ingelheim Investigational Site, Frederiksberg C
  - Lungemedicinsk Forskning, Hellerup
  - Medical Dept. B0642, Hillerød
  - Hvidovre Hospital, Hvidovre
  - Gynækologisk/obstetrisk afd., Kolding
- Finland (5):
  - Boehringer Ingelheim Investigational Site, Hyvinkää
  - Boehringer Ingelheim Investigational Site, Jyväskylä
  - Kuopion yliopistollinen sairaala, Keuhkoklinikka, Kuopio
  - Boehringer Ingelheim Investigational Site, Riihimäki
  - Boehringer Ingelheim Investigational Site, Tampere
- Netherlands (2):
  - Bosch Medicentrum, 's-Hertogenbosch
  - Dept. of Internal Medicine, Utrecht
- Norway (4):
  - Boehringer Ingelheim Investigational Site, Arendal
  - Boehringer Ingelheim Investigational Site, Jessheim
  - Boehringer Ingelheim Investigational Site, Skogn
  - Hjertelaget Research Foundation, Stavanger
- Sweden (8):
  - Medicinkliniken, Eksjö
  - Medicinkliniken, Helsingborg
  - Boehringer Ingelheim Investigational Site, Helsingborg
  - Boehringer Ingelheim Investigational Site, Munkedal
  - Boehringer Ingelheim Investigational Site, Tranås
  - Boehringer Ingelheim Investigational Site, Uddevalla
  - Samariterhemmets sjukhus, Uppsala
  - Boehringer Ingelheim Investigational Site, Vetlanda
- United Kingdom (12):
  - Boehringer Ingelheim Investigational Site, Atherstone
  - Boehringer Ingelheim Investigational Site, Barry
  - Dept. of Diabetes, Birmingham
  - Department of Respiratory Medicine, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - Finance Office (Research Unit), Newcastle upon Tyne
  - Northampton General Hospital, Northampton
  - Boehringer Ingelheim Investigational Site, Northampton
  - Diabetes Centre,, Nuneaton
  - Lucille Packard Children's Health Services at Stanford, Palo Alto
  - Boehringer Ingelheim Investigational Site, Pont-y-clun
  - Diabetes Centre, Rugby

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786